CLINICAL TRIAL: NCT05201833
Title: Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI)- a Longitudinal Biomarker Study
Brief Title: TRACK-TBI Longitudinal Biomarker Study
Acronym: TRACK-BIO
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Football League (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 834982; U01NS114140 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biofluids that will be collected and stored include serum, plasma, DNA and RNA. Samples will be banked at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Telephone Assessment Battery: TRACK-TBI participants may complete up to three annual telephone calls to assess outcome status. These assessments will determine eligibility for the in-person study visit.
  Interventions: Behavioral: Telephone Outcome Assessment
- Comprehensive Assessment Battery (CAB): Participants who demonstrate decision-making capacity will be asked to complete the Comprehensive Assessment Battery (CAB). The CAB in-person is comprised of measures of cognition (i.e. attention, memory, information processing speed, executive functions), mood (i.e., depression, anxiety), social participation, subjective well-being, post-traumatic stress, interviews, global functional status measures, and a COVID-19 questionnaire.
  Interventions: Behavioral: Telephone Outcome Assessment; Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Procedure: Blood Draw
- Abbreviated Assessment Battery (AAB): Participants who do not have decision-making capacity will be asked to complete a modified assessment battery, called the Abbreviated Assessment Battery (AAB). The AAB in-person assessment will administer the Speech Intelligibility, GOAT, and CAP and/or CRS-R to study participants.
  Interventions: Behavioral: Telephone Outcome Assessment; Behavioral: In-Person Outcome Assessment; Procedure: 3T Magnetic Resonance Imaging (MRI); Procedure: Blood Draw

INTERVENTIONS:
Behavioral: Telephone Outcome Assessment — Assessments will be administered over the telephone to evaluate participant outcome status
Behavioral: In-Person Outcome Assessment — Assessments will be administered to evaluate participant outcome status
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB)
Procedure: 3T Magnetic Resonance Imaging (MRI) — Participants will be asked to complete a 3T MRI
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB)
Procedure: Blood Draw — Blood Draw for Plasma, DNA, Serum, RNA
  Groups: Abbreviated Assessment Battery (AAB); Comprehensive Assessment Battery (CAB)

SUMMARY:
The overarching goal of this study is to improve understanding of the long-range natural history of TBI by extending follow-up of a previously enrolled cohort (TRACK-TBI) beyond the first 12 months after injury.

DETAILED DESCRIPTION:
This longitudinal observational study is part of the Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) initiative, a multi-institutional project designed to characterize the acute and longer-term clinical, neuroimaging, and blood biomarker features of TBI. TRACK-TBI enrolled TBI patients at 18 Level 1 Trauma Centers in the US, across the age and injury spectrum. This study will extend the follow-up period for TRACK-TBI participants. The extensive clinical, imaging, and biomarker data that has already been collected in these TRACK-TBI participants, in combination with the extended longitudinal data, will allow for the identification of risk factors, co-morbidities, and prognostic biomarkers of TBI. Consequently, the extension of study follow-up will help to determine negative neurological and psychological outcomes of individuals who experienced a TBI compared to healthy and orthopedic controls.

TBI is a complex disease process, in which diverse injury subtypes and multiple molecular mechanisms overlap. There is a need to identify and measure these subtypes, in order to develop precision medicine approaches where specific pathobiological processes are targeted by mechanistically appropriate therapies. The absence of validated biomarkers in the neurotrauma field is a barrier to drug development in this area, and there are currently no disease-modifying therapies that limit the burden of TBI. Biomarkers specific for injury mechanisms should be identified to select participants for clinical trials of targeted therapies (prognostic biomarkers), as well as to confirm target engagement and biological efficacy (pharmacodynamic biomarkers).

Traumatic axonal injury (TAI) is a common pathologic consequence of TBI, and underlies some of the most disabling consequences of injury, including cognitive and affective problems. TAI progresses for years after injury in a subset of patients, and is a key mechanism for long-term neurodegeneration after TBI. Recent breakthroughs in pre-clinical models indicate that novel therapeutic interventions, including strategies such as targeting the mitochondrial transition pore, or promoting axonal maintenance factors are effective in promoting resilience of injured axons and improving neurologic outcome after experimental TBI. Translation of such promising therapies into clinical trials will require prognostic biomarkers that can measure TAI in individual patients, so they can be selected for early phase studies of axon-protective therapies, as well pharmacodynamic biomarkers than can measure the biologic efficacy of such treatments. Currently, the best biomarker for TAI is fractional anisotropy (FA) and mean diffusivity (MD) of white matter tracts, measured using diffusion tensor imaging (DTI) MRI. This technique, while robust, is poorly suited for dynamic longitudinal assessments, and measures the end-result of axonal degeneration, rather than an early step in the neurodegenerative process. Recently, the ability to assay axonal proteins in peripheral blood has made it potentially feasible to assess of TAI rapidly, inexpensively, and longitudinally. The axonal protein that holds the most promise as a biomarker of axonal degeneration is neurofilament light chain (NF-L). This project aims to address the gaps in the existing literature regarding specific biomarkers for injury mechanisms and outcomes following TBI. Furthermore, it is likely that a sophisticated understanding of the subtypes and molecular mechanisms of TBI will be required to successfully develop therapies to treat these subtypes.

ELIGIBILITY:
Inclusion Criteria:

* LONGITUDINAL Telephone Assessment:
* Participated in TRACK-TBI,
* At least two years post injury, and
* Completed at least 1 GOSE during the TRACK-TBI follow-up assessments
* LONGITUDINAL BIOMARKER In-Person Assessment:

Must complete at least one Longitudinal Telephone Assessment and fall into one of the following groups:

* Group 1- Completed TRACK-TBI 6M MRI and are stable or improved with regard to Criteria for Establishing Decline
* Group 2- Criteria for Establishing Decline met when comparing the Telephone Assessments to the last completed TRACK-TBI assessment
* Group 3- All TRACK-TBI orthopedic controls

Ability of participant or legally authorized representative to provide informed consent

Exclusion Criteria:

* Dementia diagnosed prior to the index TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in TRACK-TBI
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | ~4-6 years post-injury
  The GOSE provides an overall measure of functional status based on information on cognition, independence, employability, and social/community participation collected via structured interview. Individuals are described by one of the eight outcome categories: Dead (1); Vegetative State (2); Lower Severe Disability (3); Upper Severe Disability (4); Lower Moderate Disability (5); Upper Moderate Disability (6); Lower Good Recovery (7) and Upper Good Recovery (8). Good Recovery is defined as a score of 7-8, Moderate Disability is defined by a score of 5-6 and Severe Disability is defined by a score of 3-4.

SECONDARY OUTCOMES:
Serum NF-L (neurofilament light chain) | ~4-6 years post-injury
  Using advanced blood-based assay platforms, levels of blood biomarkers neurofilament light chain (NF-L) will be measured to validate the utility as a biomarkers for traumatic axonal injury (TAI).

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania/Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No